CLINICAL TRIAL: NCT06974422
Title: Efficacy of Aerobic Training Using Lower Body Positive Pressure Technology on Cardiovascular Disease Risk and Peripheral Vascular Health in Patients With Type 2 Diabetes Mellitus. Randomized Controlled Study
Brief Title: Weight Off-loading Training, Cardiovascular Indices, Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ashraf Abdelaal, Principal Investigator, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNEZ070525
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Disease, Diabetes Mellitus Type 2; Peripheral Vascular Disorder Due to Diabetes Mellitus
Keywords: Exercise; Partial Weight-Bearing; Type 2 Diabetes Mellitus; Cardiovascular Disease; Ankle Brachial Index
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group-1 (group-A; 0% weight off-loading) (Active Comparator): This group (100% weight-bearing group) received three sessions per week of moderate-intensity (60-75% heart rate reserve) aerobic exercise training, for 12 weeks, 50-60 minutes' session duration (including warm-up and cool-down), on the antigravity treadmill. Participants also received regular oral anti-diabetic medications.
  Interventions: Behavioral: Full weight bearing during aerobic exercise training
- Experimental Group-2 (group-B; 25% weight off-loading) (Experimental): This group (27% weight-bearing group) received three sessions per week of moderate-intensity (60-75% heart rate reserve) aerobic exercise training, for 12 weeks, 50-60 minutes' session duration (including warm-up and cool-down), on the antigravity treadmill. Participants also received regular oral anti-diabetic medications.
  Interventions: Behavioral: Partial weight bearing during aerobic exercise training
- Control group (Group; Non-exercising group) (Other): The control group participants received the same pre- and post-study evaluations as those for the study groups A and B, but did not participate in any aerobic exercise training on the antigravity treadmill. Participants only received regular oral anti-diabetic medications.
  Interventions: Drug: Regular oral anti-diabetic medications.

INTERVENTIONS:
Behavioral: Partial weight bearing during aerobic exercise training — Partial weight bearing (25% weight support) during the moderate intensity aerobic exercise training on the antigravity treadmill
  Other Names: Antigravity treadmill aerobic exercise training; partial weight offloading during aerobic exercise training
  Arms: Experimental Group-2 (group-B; 25% weight off-loading)
Behavioral: Full weight bearing during aerobic exercise training — Full weight bearing (100% weight loading, 0% weight support) during moderate intensity aerobic exercise training on the antigravity treadmill.
  Arms: Experimental Group-1 (group-A; 0% weight off-loading)
Drug: Regular oral anti-diabetic medications. — Participants in the control group (group C) received regular oral anti-diabetic medications.
  Arms: Control group (Group; Non-exercising group)

SUMMARY:
Aims: To evaluate the effectiveness of partial weight-bearing during aerobic exercise training on cardiovascular disease risk and peripheral vascular function in patients with type 2 diabetes mellitus.

Study design: A Randomized controlled study was conducted in the outpatient rehabilitation unit.

Population: Forty-six participants (age 60 -70) with type 2 diabetes mellitus were recruited and randomly allocated into three groups: group A (100% weight-bearing; n=16), group B (75% weight-bearing; n=16), and group C (control group; n=14).

Methods: The 2 study groups A and B, received three sessions per week of moderate intensity (60-75% heart rate reserve) aerobic exercise training, for 12 weeks, 50-60 minutes session duration (including warm-up and cool-down), on the antigravity treadmill. The cardiovascular disease risk (evaluated using the Atherosclerotic cardiovascular disease risk estimator plus tool) and peripheral vascular function (presented by ankle-brachial pressure index, calculated by subdividing the ankle systolic blood pressure by the brachial systolic blood pressure) are the main study outcomes. Variables were evaluated pre-study and post-study. Ethical concepts and institutional regulations were adhered during the study. Data were described as mean and standard deviation. Paired samples t-test and one-way ANOVA were used to test within and between-subjects assumptions, respectively, considering p< 0.05 as the significance level.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) continues as a global alarming epidemic, with an increasingly growing health burden and complications across all socioeconomic levels. Type 2 diabetes mellitus (T2DM) is associated with wide peripheral vascular complications, manifested in deteriorated lower limb blood pressure and vascular endothelial dysfunction. Prevalence of peripheral vascular disorder varies with T2DM duration, ranging from 1.2% in newly discovered T2DM cases, to about 12.5% (after 18 years of T2DM affection), and reaches 20-30% in some reports.

The abnormally increased cardiovascular disease CVD (either through traditional risk factors or direct diabetes effects) is expected to continue rising alongside DM. Adequate management for DM and associated CVD risk factors is essential to ameliorate the progression of DM and CVD.

Being active is beneficial in alleviating the peripheral vascular disease burden in patients with disturbed peripheral vascular function. Supervised treadmill exercise training can improve functional performance in patients with peripheral arterial disorders. Increasing patients' activity level is a cornerstone item in patients with T2DM rehabilitation programs.

Patients may be challenged by the disease-related pathophysiological changes and treatment requirements. The hallmark of inactivity status that dominates in patients with T2DM negatively impacts their performance during weight-bearing activities. The existence of pain, peripheral vascular disturbances, abnormally increased and unequally distributed plantar stress, all limit patients' participation and compliance with the full weight-bearing training programs.

Introducing the well-controlled partial weight-bearing through the lower body positive pressure technology during exercise training programs augments patients' active participation, minimizes weight-bearing related musculoskeletal limitations, while maintaining normal locomotion dynamics and training-related physiological responses.

Conflicts arise regarding the benefits of full and partial weight-bearing exercise training for patients with T2DM. Previous studies investigated the effects of modulating the weight-bearing status during aerobic exercise training on different health aspects and concluded conflicting results. Quite recently published studies reported the safety and efficacy of the partial weight-bearing AET training in improving the T2DM-related musculoskeletal constraints.

To our knowledge, this study is the first to investigate the effects of partial weight bearing during AET on cardiovascular variables in patients with T2DM. The objectives of this study were to evaluate the effectiveness of partial weight off-loading during aerobic exercise training, using the antigravity treadmill, on the cardiovascular disease risk and the peripheral vascular health (presented by the ankle-brachial pressure index) in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients with 0.6< ankle brachial index ≤ 0.9, treated only with oral hypoglycemic medications (Biguanide or Sulfonylureas + Biguanide), oral anti-diabetic drugs combination, with stable pharmacological treatment for at least 3 months before the study.
* Cognitively competent patients, able to walk independently with or without walking aids, assuming a Sedentary lifestyle (less than 30 minutes daily activity) during the last 6 months.
* Type 2 diabetes mellitus for more than 10 years, with glycosylated hemoglobin (HbA1c% %) level more than 7%, and fasting glucose level more than 7.0 mmol/L.
* Age range from 60 to 70 years, with normal/ accepted nutritional status (Mini Nutritional Assessment score more than 11).

Exclusion Criteria:

* The following condition resulted in the exclusion of the patients from the study at the initial screening stage:
* Patients with Type 1 diabetes, younger than 60 or older than 70 years.
* Participation in any previous training program or diet regimen within the last 6 months.
* Patients with disturbed nutritional status (Mini Nutritional Assessment score less than 11).
* Serious musculoskeletal or cardiopulmonary disorders that can affect patient safety or the study results.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in the cardiovascular disease risk at 12-week. | From enrollment to the end of treatment at 12 weeks.
  The cardiovascular disease risk was evaluated using the Atherosclerotic cardiovascular disease risk estimator plus tool, and was evaluated pre-study and at 12 weeks (end of the study).
Change in the peripheral vascular function at 12-week. | From enrollment to the end of treatment at 12 weeks.
  The peripheral vascular function (presented by ankle-brachial pressure index) was calculated by dividing the ankle systolic blood pressure by the brachial systolic blood pressure, and was evaluated pre-study and at 12 weeks (end of the study).

CONTACTS AND LOCATIONS:
Overall Officials: ASHRAF AM ABDELAAL, Ph.D., Principal Investigator — Associate Professor
Locations (1):
- Umm Al-Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
For privacy reasons, data can not be exposed until results' publication. Data summary will be confidentially provided upon request under limited situations.